CLINICAL TRIAL: NCT03844425
Title: Microbial Colonisation On Vacuum-Formed Retainers With Different Surface Roughness As Constructed On Conventional Models And Three Dimensional (3D) Reconstructed Models
Brief Title: Microbial Colonisation On Vacuum-Formed Retainers Constructed On Conventional Models And Three Dimensional (3D) Reconstructed Models
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Malaya (Other)
Responsible Party: Principal Investigator, Dr Wan Nurazreena Wan Hassan, Associate Professor, Department Of Paediatric Dentistry & Orthodontics, Faculty Of Dentistry, University of Malaya
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: DGD_170002
Record Dates: First submitted 2019-02-14; First posted 2019-02-18 (Actual); Last update posted 2021-05-26 (Actual); Status verified 2021-05

CONDITIONS: Orthodontic Appliance Complication
Keywords: Orthodontic Retainers; Printing, Three-Dimensional; Colony Count, Microbial

STUDY DESIGN:
Who Masked: Investigator
Masking Description: Investigator will be masked with the randomization sequance & allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Conventional Vacuum-Formed Retainers (Active Comparator): Vacuum-formed retainers constructed on conventional stone models.
  Interventions: Device: Conventional VFR
- Vacuum-Formed Retainers From SLA (Experimental): Vacuum-formed retainers constructed on 3D reconstructed models using stereolitography (SLA) technique.
  Interventions: Device: VFR from SLA
- Vacuum-Formed Retainers From FDM (Experimental): Vacuum-formed retainers constructed on 3D reconstructed models using fused deposition modeling technique (FDM).
  Interventions: Device: VFR from FDM

INTERVENTIONS:
Device: Conventional VFR — Conventional retainers
  Arms: Conventional Vacuum-Formed Retainers
Device: VFR from SLA — SLA has better finishing compared to FDM but it is more expensive.
  Arms: Vacuum-Formed Retainers From SLA
Device: VFR from FDM — FDM has poorer finishing compared to SLA but it is cheaper.
  Arms: Vacuum-Formed Retainers From FDM

SUMMARY:
Vacuum-formed retainers are clear or transparent retainers, that hold the teeth in the new position after active orthodontic treatment. These custom made appliances are becoming popular these days due to the aesthetics value among patients.

Vacuum-formed retainers can be made through a process that softens the clear plastic and vacuumed to follow the shape of the dental model before it cools off and hardens again. These dental models can be made from conventional method or through a 3D reconstruction process. Recently, it was found that there is no difference in terms of stability of the teeth and oral health related quality of life of the patients wearing vacuum-formed retainers constructed on either types of models.

Physically, the surface roughness of the retainers appear different because the conventional models and 3D printed models are constructed in a different manner.

Our interest is to determine whether the difference in surface roughness would affect microbial colonisation which can eventually affect the oral health.

So this study aims to find the association between microbial colonisation and surface roughness of vacuum-formed retainers constructed on conventional models and also 3D reconstructed models.

DETAILED DESCRIPTION:
RATIONALE OF STUDY

The vacuum-formed retainers are widely preferred today but there is limited research on the effects of the retainers on microbial colonisation, which can have an impact on the oral health. There is possibility that a rough surface finishing of the vacuum-formed retainers may lead to increased microbial colonisation. Therefore, there is a need for us to investigate if the vacuum formed retainers made on 3D reconstructed models may produce increased surface roughness which then can lead to increased microbial colonisation and later impacts the oral health.

Primary Objective :

1. To determine the association between different surface roughness of vacuum- formed retainers and microbial colonisation.

Secondary Objectives :

1. To compare the surface roughness of vacuum-formed retainers constructed on conventional models and 3D reconstructed models.
2. To compare the microbial colonisation on vacuum-formed retainers with different roughness as constructed on conventional models and 3D reconstructed models.
3. To compare the microbial colonisation between upper and lower vacuum-formed retainers with different surface roughness.
4. To compare the microbial colonisation on vacuum-formed retainers with different surface roughness between full time wear and part time wear.

SAMPLE SIZE CALCULATION

Sample size calculation is done based on a type 1 error frequency of 5% and the power of the statistical test is set at 80%. This is based on a study done by Farhadian et al, 2016 on Streptococcus colonisation on orthodontic retainers. The total number of participant needed for the trial was 27 with a minimum of 9 participants per group. With an anticipated 20% drop outs, a total number of 36 patients will be recruited.

Methodology

Patients who are currently undergoing fixed appliance treatment at Faculty of Dentistry, University of Malaya will be screened for their progress of treatment and whether they are ready for debond. During screening, patients who fit the inclusion and exclusion criteria will be selected and given a patient information sheet and a detailed explanation of the clinical trial. Voluntarily participant will then be recruited into this study and informed consent will be obtained. A total number of 36 participants will be recruited for this clinical trial.

Participants will be drawing lots to obtain their study number. Then, the orthodontic resident will have to check the group allocation with the orthodontic consultant.

During the first appointment, debond procedure will be done according to the standard protocol. Three sets of impression will be taken for the construction of study model, construction of the standard retainers and also for the research purpose. The standard retainers will then be issued on the same day of debond (T0). Participants will be instructed to wear the retainers full time except during brushing, cleaning of the appliance and during meals.

Participants will be reviewed one week post debond (T1). During this appointment, the standard retainers will be taken and kept by the orthodontic resident. The first interventional retainers will be issued and participants are advised to wear the retainers full time / 24 hours except during meals, brushing and cleaning of the appliance. Participants will be given a new retainer box to keep their retainers as well as a new toothbrush for cleaning their appliance. A pamphlet that contains detailed information on the care of retainers will also be provided to every participant. Participants will be reminded regularly to wear their retainers full time / 24 hours for three months.

Participants will be reviewed again 3 months post debond (T2). During this appointment, the first interventional retainers will be taken and kept by the orthodontic resident. Then the second interventional retainers will be issued and participants are advised to wear the retainers for 10 hours only. Participants will also be given a new retainer box to keep their retainers as well as a new toothbrush for cleaning their appliance. Analysis of the first interventional retainers will then be carried out. Participants will also be reminded regularly to wear their retainers for 10 hours only for 3 months.

Participants will be reviewed again 6 months post debond (T3). During this appointment, the second interventional retainers will be taken and kept by the orthodontic resident. Then the standard retainers will be issued back and participants are advised to continue wearing the retainers for 10 hours only. Analysis of the second interventional retainers will then be carried out.

STATISTICAL ANALYSIS

Statistical Analysis will be done using SPSS software version 21. P < 0.05 will be set as the level of significance.

i. One way analysis of variance (ANOVA) will be used to compare the surface roughness and microbial colonization on vacuum-formed retainers constructed on conventional models and 3D reconstructed models.

ii. Paired Sample T-Test will be used to compare the microbial colonization between the upper and lower vacuum-formed retainers with different surface roughness as well as between full time wear and part time wear.

iii. Correlation will be used to determine the association between surface roughness of vacuum-formed retainers and microbial colonization.

ELIGIBILITY:
Inclusion Criteria:

i. Fixed appliance on upper and lower arches ii. About to debond iii. Planned for vacuum-formed retainers for retention iv. Non smoking patients v. No systemic disease

Exclusion Criteria:

i. Undergoing sectional fixed appliance / single arch treatment ii. Indicated for double retention regime with bonded retainers iii. Patient with smoking habit iv. Any systemic disease that may affect the salivary flow v. History of use of antimicrobial mouthwash less than 1 month prior to debond

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2019-12-02 (Actual); Primary Completion 2021-04-10 (Actual); Study Completion 2021-04-10 (Actual)

PRIMARY OUTCOMES:
Microbial Colonisation On Vacuum-Formed Retainers | 6 months
  Microbial colony count on the vacuum-formed retainers constructed on conventional models & 3D reconstructed models.
  The vacuum-formed retainers that are collected from the patients will be placed in BHI media and then undergo the process of sonication, which will produce the bacteria suspension. This bacteria suspension will then be cultured in an agar plate with BHI media and incubated for 18 - 24 hours. The total colony per count will then be counted and recorded.

SECONDARY OUTCOMES:
Surface Roughness Of Vacuum-Formed Retainers | 6 months
  Surface roughness values of vacuum-formed retainers constructed on conventional models & 3D reconstructed models.
  The surface roughness of the vacuum-formed retainers will be measured using Alicona 3D Surface Management System. Vacuum-formed retainers which are new and used by patient (after disinfection) will be placed for surface roughness assessment under the microscope and the value which is measured as Ra (profile roughness parameter) will be recorded.

OTHER OUTCOMES:
Patient's Compliance In Wearing Vacuum-Formed Retainers | 6 months
  Patients's compliance in wearing vacuum-formed retainers as instructed.
  Patient's compliance will be measured using a global rating scale that asked if they wore the VFR 24 hours or 10 hours per day as instructed. If the patient admitted to wear the retainers more than 24 hours or 10 hours daily as instructed, the patient is considered to be compliant.

CONTACTS AND LOCATIONS:
Locations (1):
- Postgraduate Orthodontic Clinic, Faculty Of Dentistry, University Of Malaya, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dawes C, Watanabe S, Biglow-Lecomte P, Dibdin GH. Estimation of the velocity of the salivary film at some different locations in the mouth. J Dent Res. 1989 Nov;68(11):1479-82. doi: 10.1177/00220345890680110201. PMID 2531176
- [Background] Dawes C. Salivary flow patterns and the health of hard and soft oral tissues. J Am Dent Assoc. 2008 May;139 Suppl:18S-24S. doi: 10.14219/jada.archive.2008.0351. PMID 18460676
- [Background] Dietrich CA, Ender A, Baumgartner S, Mehl A. A validation study of reconstructed rapid prototyping models produced by two technologies. Angle Orthod. 2017 Sep;87(5):782-787. doi: 10.2319/01091-727.1. Epub 2017 May 1. PMID 28459285
- [Background] Hazeveld A, Huddleston Slater JJ, Ren Y. Accuracy and reproducibility of dental replica models reconstructed by different rapid prototyping techniques. Am J Orthod Dentofacial Orthop. 2014 Jan;145(1):108-15. doi: 10.1016/j.ajodo.2013.05.011. PMID 24373661
- [Background] Hibino K, Wong RW, Hagg U, Samaranayake LP. The effects of orthodontic appliances on Candida in the human mouth. Int J Paediatr Dent. 2009 Sep;19(5):301-8. doi: 10.1111/j.1365-263X.2009.00988.x. Epub 2009 Apr 16. PMID 19486368
- [Background] Hichens L, Rowland H, Williams A, Hollinghurst S, Ewings P, Clark S, Ireland A, Sandy J. Cost-effectiveness and patient satisfaction: Hawley and vacuum-formed retainers. Eur J Orthod. 2007 Aug;29(4):372-8. doi: 10.1093/ejo/cjm039. PMID 17702797
- [Background] Kasparova M, Grafova L, Dvorak P, Dostalova T, Prochazka A, Eliasova H, Prusa J, Kakawand S. Possibility of reconstruction of dental plaster cast from 3D digital study models. Biomed Eng Online. 2013 May 31;12:49. doi: 10.1186/1475-925X-12-49. PMID 23721330
- [Background] Keating AP, Knox J, Bibb R, Zhurov AI. A comparison of plaster, digital and reconstructed study model accuracy. J Orthod. 2008 Sep;35(3):191-201; discussion 175. doi: 10.1179/146531207225022626. PMID 18809782
- [Background] Kim GB, Lee S, Kim H, Yang DH, Kim YH, Kyung YS, Kim CS, Choi SH, Kim BJ, Ha H, Kwon SU, Kim N. Three-Dimensional Printing: Basic Principles and Applications in Medicine and Radiology. Korean J Radiol. 2016 Mar-Apr;17(2):182-97. doi: 10.3348/kjr.2016.17.2.182. Epub 2016 Mar 2. PMID 26957903
- [Background] Low B, Lee W, Seneviratne CJ, Samaranayake LP, Hagg U. Ultrastructure and morphology of biofilms on thermoplastic orthodontic appliances in 'fast' and 'slow' plaque formers. Eur J Orthod. 2011 Oct;33(5):577-83. doi: 10.1093/ejo/cjq126. Epub 2010 Dec 27. PMID 21187528
- [Background] Mamai-Homata E, Koletsi-Kounari H, Margaritis V. Gender differences in oral health status and behavior of Greek dental students: A meta-analysis of 1981, 2000, and 2010 data. J Int Soc Prev Community Dent. 2016 Jan-Feb;6(1):60-8. doi: 10.4103/2231-0762.175411. PMID 27011935
- [Background] Marsh PD. The role of microbiology in models of dental caries. Adv Dent Res. 1995 Nov;9(3):244-54; discussion 255-69. doi: 10.1177/08959374950090030901. PMID 8615947
- [Background] Quirynen M, Marechal M, Busscher HJ, Weerkamp AH, Darius PL, van Steenberghe D. The influence of surface free energy and surface roughness on early plaque formation. An in vivo study in man. J Clin Periodontol. 1990 Mar;17(3):138-44. doi: 10.1111/j.1600-051x.1990.tb01077.x. PMID 2319000
- [Background] Thickett E, Power S. A randomized clinical trial of thermoplastic retainer wear. Eur J Orthod. 2010 Feb;32(1):1-5. doi: 10.1093/ejo/cjp061. Epub 2009 Oct 14. PMID 19828592
- [Background] Turkoz C, Canigur Bavbek N, Kale Varlik S, Akca G. Influence of thermoplastic retainers on Streptococcus mutans and Lactobacillus adhesion. Am J Orthod Dentofacial Orthop. 2012 May;141(5):598-603. doi: 10.1016/j.ajodo.2011.11.021. PMID 22554754
- [Background] Wan Hassan WN, Yusoff Y, Mardi NA. Comparison of reconstructed rapid prototyping models produced by 3-dimensional printing and conventional stone models with different degrees of crowding. Am J Orthod Dentofacial Orthop. 2017 Jan;151(1):209-218. doi: 10.1016/j.ajodo.2016.08.019. PMID 28024776
- [Background] Yitschaky O, Katorza A, Zini A, Yitschaky M, Zadik Y. Acrylic orthodontic retainer is not a risk factor for focal Candida colonization in young healthy patients: a pilot study. Oral Surg Oral Med Oral Pathol Oral Radiol. 2016 Jan;121(1):39-42. doi: 10.1016/j.oooo.2015.10.001. Epub 2015 Oct 22. PMID 26679358
- [Derived] Belayutham S, Wan Hassan WN, Razak FA, Mohd Tahir NNZ. Microbial adherence on vacuum-formed retainers with different surface roughness as constructed from conventional stone models and 3D printed models: a randomized controlled clinical trial. Clin Oral Investig. 2023 Jun;27(6):3245-3259. doi: 10.1007/s00784-023-04940-4. Epub 2023 Mar 22. PMID 36947263